CLINICAL TRIAL: NCT05510271
Title: The Effect of White Noise and Therapeutic Touch on Pain in Newborn Heel Blood Collection
Brief Title: Pain in Newborn Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: MSc Reyhan YALÇIN (Unknown); MSc Meral Güven (Unknown)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ATA.0.01.00/124
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Infant, Newborn, Disease; Pain, Acute
MeSH Terms: conditions — Disease; Acute Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White Noise (Experimental)
  Interventions: Other: White Noise
- Yakson touch (Experimental)
  Interventions: Other: Yakson Touch
- Control (No Intervention)

INTERVENTIONS:
Other: White Noise — Orhan OSMAN's song "Don't Let Your Baby Cry-2" from the "Kolik" album was used.
  Arms: White Noise
Other: Yakson Touch — In order to transfer the Ki energy to the baby, he took a deep breath and gathered the universal energy in his palms, intending the baby's well-being and healing. The researcher applied the Yakson touch by covering the abdomen and chest of the newborn with his right hand (dominant hand) while the newborn was in the supine position, and supported the baby's back and hips with his left hand.
  Arms: Yakson touch

SUMMARY:
This study was conducted to evaluate the effect of white noise and therapeutic touch on pain in newborn heel blood collection.Questions including the sex of the newborns, postnatal age, gestational age, birth weight, height, head and chest circumference, feeding style, nutritional status in the last half hour, and previous heel blood collection were collected with the "Information Form".The Newborn Infant Pain Scale (NIPS) was used to evaluate the pain levels of newborns.

ELIGIBILITY:
Inclusion Criteria:

* gestational week 37 and above,
* fasting time < 1 hour,
* without comorbidity and congenital anomalies,
* not receiving oxygen or mechanical respiratory support,
* no analgesic sedation before the procedure
* neonates with stable physiological findings before the procedure

Exclusion Criteria:

• newborns whose heel blood cannot be taken at once

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The Newborn Infant Pain Scale (NIPS) | 12 week
  The Newborn Infant Pain Scale (NIPS) was used. NIPS: Scale Lawrence et al. (1993) was developed to evaluate the behavioral and physiological pain responses of preterm and term infants. The scale consists of five behavioral factors (facial expression, crying, arousal, arm and leg movements) and one physiological (breathing pattern) factor. The crying factor is given 0-1-2 points, the other factors are given 0-1 points, and the total score is between 0-7. A high score indicates greater severity of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No